CLINICAL TRIAL: NCT03219333
Title: A Single-arm, Open-label, Multicenter Study of Enfortumab Vedotin (ASG-22CE) for Treatment of Patients With Locally Advanced or Metastatic Urothelial Cancer Who Previously Received Immune Checkpoint Inhibitor (CPI) Therapy
Brief Title: A Study of Enfortumab Vedotin for Patients With Locally Advanced or Metastatic Urothelial Bladder Cancer
Acronym: EV-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN22E-001
Expanded Access: NCT04136808 (Approved for marketing)
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urologic Neoplasms; Renal Pelvis Neoplasms; Urothelial Cancer; Ureteral Neoplasms; Urethral Neoplasms
Keywords: Enfortumab vedotin; Metastatic Urothelial Cancer; ASG-22CE; Locally Advanced Urothelial Cancer; Antibody-Drug Conjugate; Nectin-4; Platinum-naïve; Cisplatin-ineligible; Antineoplastic Agents; Drug Therapy; ASG-22ME
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urologic Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: single-arm, open-label, multi-cohort, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enfortumab vedotin (Experimental): Enfortumab vedotin on days 1, 8 and 15 every 28 days
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Intravenous (IV) infusion on days 1, 8 and 15 every 28 days
  Other Names: ASG-22CE; ASG-22ME

SUMMARY:
This is a study that will test how an experimental drug (enfortumab vedotin) affects patients with cancer of the urinary system (urothelial cancer). This type of cancer includes cancer of the bladder, renal pelvis, ureter or urethra that has spread to nearby tissues or to other areas of the body.

This clinical trial will enroll patients who were previously treated with a kind of anticancer drug called an immune checkpoint inhibitor (CPI). Some CPIs have been approved for the treatment of urothelial cancer.

This study will test if the cancer shrinks with treatment. This study will also look at the side effects of the drug. A side effect is a response to a drug that is not part of the treatment effect.

Patients who sign up for this trial must also fall into one of these categories:

* Patients have already received treatment with platinum-containing chemotherapy
* Patients have never received platinum-containing treatment and are not eligible for treatment with cisplatin.

DETAILED DESCRIPTION:
Japan Pharmaceuticals and Medical Devices Agency (PMDA) has approved enfortumab vedotin (Padcev) for the treatment of advanced urothelial cancer. The study will continue as a post marketing study in Japan.

This study will examine the safety and anticancer activity of enfortumab vedotin given intravenously to patients with locally advanced or metastatic urothelial cancer who previously received a CPI and either previously received platinum-containing chemotherapy (Cohort 1) or are platinum-naïve and cisplatin-ineligible (Cohort 2). Patients who received platinum in the adjuvant/neoadjuvant setting and did not progress within 12 months of completion will be considered platinum-naïve. Approximately 100 patients are expected to be enrolled in each cohort. The primary goal of the study is to determine the confirmed ORR of enfortumab vedotin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented urothelial carcinoma (squamous differentiation or mixed cell types allowed).
* Metastatic disease or locally advanced disease that is not resectable.
* Must have received prior treatment with a CPI in the locally advanced or metastatic urothelial cancer setting. A CPI is defined as a programmed cell death protein 1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitor. Patients who received CPI therapy in the neoadjuvant/adjuvant setting and had recurrent or progressive disease either during therapy or within 3 months of therapy completion are eligible.
* Must either have prior treatment with platinum-containing chemotherapy (Cohort 1) or be platinum-naïve and ineligible for treatment with cisplatin at time of enrollment (Cohort 2).
* Must have had progression or recurrence of urothelial cancer during or following receipt of most recent therapy.
* Tumor tissue samples must be available for submission to the sponsor prior to study treatment.
* Must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1).
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤1 for Cohort 1 or ≤2 for Cohort 2.
* Anticipated life expectancy of ≥3 months as assessed by the investigator.

Exclusion Criteria:

* Ongoing sensory or motor neuropathy Grade ≥2.
* Active central nervous system (CNS) metastases.
* Immunotherapy related myocarditis, colitis, uveitis, or pneumonitis.
* Prior enrollment in an enfortumab vedotin study or prior treatment with other monomethyl auristatin E (MMAE)-based antibody-drug conjugates (ADCs).
* Uncontrolled tumor-related pain or impending spinal cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Trowbridge, MD, PhD, Study Director — Seagen Inc.
Locations (81):
- United States (54):
  - Alaska Urological Institute, Anchorage, Alaska
  - Arizona Oncology Associates, PC - HAL, Goodyear, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Keck Medical Center / University of Southern California, Los Angeles, California
  - Keck Medical Center / Newport Beach, Newport Beach, California
  - Kaiser Permanente Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center University of California Irvine, Orange, California
  - University of California Irvine - Newport, Orange, California
  - Kaiser Permanente Roseville, Roseville, California
  - University of California Davis, Sacramento, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Kaiser Permanente San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Kaiser Permanente South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Center Northern California, Vallejo, California
  - Kaiser Permanente Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Ocala Oncology Center, Ocala, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Washington University in St Louis, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - New York University (NYU) Cancer Institute, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center / University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC)/Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
- Site FR33001, Villejuif-Cedex-France, France
- Germany (2):
  - Site DE49004, Münster
  - Site DE49001, Tübingen
- Italy (2):
  - Site IT39001, Milan
  - Site IT39003, Terni
- Japan (12):
  - Site JP81001, Hirosaki, Aomori
  - Site JP81004, Tsukuba, Ibaraki
  - Site JP81002, Morioka, Iwate
  - Site JP81003, Nigata, Niigata
  - Site JP81008, Sayama, Osaka
  - Site JP81006, Shinjuku-ku, Tokyo
  - Site JP81009, Ube, Yamaguchi
  - Site JP81005, Chiba
  - Site JP81011, Fukuoka
  - Site JP81012, Fukuoka
  - Site JP81007, Osaka
  - Site JP81010, Tokushima
- Site NL31001, Amsterdam, Netherlands
- South Korea (5):
  - Site KR82005, Daejeon
  - Site KR82003, Seongnam-si
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82004, Seoul
- Spain (4):
  - Site ES34002, Barcelona
  - Site ES34005, Barcelona
  - Site ES34003, Santander
  - Site ES34004, Seville

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McGregor B, O'Donnell PH, Balar A, Petrylak D, Rosenberg J, Yu EY, Quinn DI, Heath EI, Campbell M, Hepp Z, McKay C, Steinberg J, Regnault A, Mazerolle F, Galsky MD. Health-related Quality of Life of Patients with Locally Advanced or Metastatic Urothelial Cancer Treated with Enfortumab Vedotin after Platinum and PD-1/PD-L1 Inhibitor Therapy: Results from Cohort 1 of the Phase 2 EV-201 Clinical Trial. Eur Urol. 2022 May;81(5):515-522. doi: 10.1016/j.eururo.2022.01.032. Epub 2022 Feb 12. PMID 35168844
- [Derived] Yu EY, Petrylak DP, O'Donnell PH, Lee JL, van der Heijden MS, Loriot Y, Stein MN, Necchi A, Kojima T, Harrison MR, Hoon Park S, Quinn DI, Heath EI, Rosenberg JE, Steinberg J, Liang SY, Trowbridge J, Campbell M, McGregor B, Balar AV. Enfortumab vedotin after PD-1 or PD-L1 inhibitors in cisplatin-ineligible patients with advanced urothelial carcinoma (EV-201): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):872-882. doi: 10.1016/S1470-2045(21)00094-2. Epub 2021 May 12. PMID 33991512
- [Derived] Rosenberg JE, O'Donnell PH, Balar AV, McGregor BA, Heath EI, Yu EY, Galsky MD, Hahn NM, Gartner EM, Pinelli JM, Liang SY, Melhem-Bertrandt A, Petrylak DP. Pivotal Trial of Enfortumab Vedotin in Urothelial Carcinoma After Platinum and Anti-Programmed Death 1/Programmed Death Ligand 1 Therapy. J Clin Oncol. 2019 Oct 10;37(29):2592-2600. doi: 10.1200/JCO.19.01140. Epub 2019 Jul 29. PMID 31356140

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants with locally advanced or metastatic urothelial cancer who have previously received systemic therapy with a programmed cell death protein-1/programmed death-ligand 1 (PD-1/PD-L1) inhibitor and met inclusion criteria and none of the exclusion criteria were enrolled in the study.
Groups:
- Enfortumab Vedotin - Cohort 1: Participants in Cohort 1 had received prior treatment with platinum-containing chemotherapy. Enfortumab vedotin, at a dose of 1.25 mg/kg, was administered to participants as an IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
- Enfortumab Vedotin - Cohort 2: Participants in Cohort 2 had received no platinum-containing chemotherapy were ineligible for treatment with cisplatin at the time of enrollment. Enfortumab vedotin, at a dose of 1.25 mg/kg, was administered to participants as an IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Started | 128 | 91
Treated | 125 | 89
Completed | 0 | 0
Not Completed | 128 | 91
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 104 | 72
Not completed — Study closed in 2023,as all milestones reached, majority of participants completed 5 years follow-up | 12 | 12
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of enfortumab vedotin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2 | Total
Number analyzed (Participants) | 125 | 89 | 214
Age, Continuous [Median (Full Range); unit: Years] | 69.0 [40 to 84] | 75.0 [49 to 90] | 72.0 [40 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 23 | 60
  Male | 88 | 66 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 118 | 83 | 201
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 20 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 106 | 62 | 168
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 117 | 57 | 174
  Europe | 0 | 14 | 14
  East Asia | 8 | 18 | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was used to assess participants disease progression, and ability to carry out daily living activities. 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0 | 40 | 37 | 77
    1 | 85 | 41 | 126
    2 | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). CR is defined as disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Cohort 1: median follow-up time: 10.15 months (range 0.49, 16.46); Cohort 2: median follow up time: 13.4 months (range 0.33 to 29.27)
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Percentage of Participants | 44 [35.1 to 53.2] | 51.7 [40.8 to 62.4]

2. Secondary Outcome: Duration of Objective Response (DOR) Per BICR
Description: The time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of progressive disease (PD) or to death due to any cause, whichever comes first. CR is defined as disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. The appearance of one or more new lesions is also considered progression. DOR was analyzed using Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 55 | 46
Months | 7.6 [6.34 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events. | 10.9 [5.78 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events.

3. Secondary Outcome: Progression-Free Survival (PFS) Per BICR
Description: The time from start of study treatment to first documentation of objective tumor progression (PD per RECIST 1.1), or to death due to any cause, whichever comes first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. The appearance of one or more new lesions is also considered progression.
Time Frame: as for outcome 1
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Months | 5.8 [4.93 to 7.46] | 5.8 [5.03 to 8.28]

4. Secondary Outcome: ORR Per Investigator Assessment
Description: ORR was defined as the percentage of participants with confirmed CR or PR according to RECIST 1.1. CR is defined as disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Percentage of Participants | 39 [30.6 to 48.3] | 50.6 [39.8 to 61.3]

5. Secondary Outcome: DOR Per Investigator Assessment
Description: CR is defined as disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. The appearance of one or more new lesions is also considered progression.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 49 | 45
Months | 7.9 [5.95 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events. | 10.7 [5.85 to 16.59]

6. Secondary Outcome: PFS Per Investigator Assessment
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Months | 5.8 [4.93 to 7.46] | 7.2 [5.42 to 7.69]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities (Hematology)
Description: A treatment-emergent laboratory abnormality is a value increases or decrease by 1 toxicity grade after the first study dose. Abnormalities were graded based on National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 - Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: The median duration of treatment was 4.60 months for Cohort 1 [range: 0.5, 29.4 months] and 5.98 months for Cohort 2 [range: 0.3, 24.6 months]
Population: Safety Analysis set. Here 'Number Analyzed' for each laboratory parameter is based on the number of participants who received at least one dose of enfortumab vedotin and have a baseline and post-baseline laboratory value.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Participants
  Hemoglobin decreased (all grades): number analyzed (Participants) | 122 | 88
  Hemoglobin decreased (all grades) | 52 | 39
  Hemoglobin decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Hemoglobin decreased (grade 3-4) | 12 | 4
  Leukocytes decreased (all grades): number analyzed (Participants) | 122 | 88
  Leukocytes decreased (all grades) | 33 | 28
  Leukocytes decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Leukocytes decreased (grade 3-4) | 5 | 4
  Lymphocytes decreased (all grades): number analyzed (Participants) | 122 | 88
  Lymphocytes decreased (all grades) | 55 | 61
  Lymphocytes decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Lymphocytes decreased (grade 3-4) | 12 | 13
  Lymphocytes increased (all grades): number analyzed (Participants) | 125 | 88
  Lymphocytes increased (all grades) | 0 | 1
  Lymphocytes increased (grade 3-4) | 0 | 0
  Neutrophils decreased (all grades): number analyzed (Participants) | 122 | 88
  Neutrophils decreased (all grades) | 28 | 27
  Neutrophils decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Neutrophils decreased (grade 3-4) | 7 | 8
  Platelets decreased (all grades): number analyzed (Participants) | 121 | 88
  Platelets decreased (all grades) | 39 | 20
  Platelets decreased (grade 3-4) | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities (Serum Chemistry)
Description: A treatment-emergent laboratory abnormality is a value increases or decrease by 1 toxicity grade after the first study dose. Abnormalities were graded based NCI CTCAE version 4.03 - Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: The median duration of treatment was 4.60 months for Cohort 1 [full range: 0.5, 29.4 months] and 5.98 months for Cohort 2 [full range: 0.3, 24.6 months]
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Participants
  Alanine aminotransferase increased (all grades): number analyzed (Participants) | 122 | 88
  Alanine aminotransferase increased (all grades) | 34 | 26
  Alanine aminotransferase increased (grade 3-4): number analyzed (Participants) | 122 | 89
  Alanine aminotransferase increased (grade 3-4) | 1 | 0
  Albumin decreased (all grades): number analyzed (Participants) | 122 | 88
  Albumin decreased (all grades) | 38 | 16
  Albumin decreased (grade 3-4): number analyzed (Participants) | 122 | 89
  Albumin decreased (grade 3-4) | 1 | 0
  Alkaline phosphatase increased (all grades): number analyzed (Participants) | 122 | 88
  Alkaline phosphatase increased (all grades) | 21 | 12
  Alkaline phosphatase increased (grade 3-4): number analyzed (Participants) | 122 | 88
  Alkaline phosphatase increased (grade 3-4) | 1 | 0
  Aspartate aminotransferase increased (all grades): number analyzed (Participants) | 121 | 88
  Aspartate aminotransferase increased (all grades) | 79 | 52
  Aspartate aminotransferase increased (grade 3-4): number analyzed (Participants) | 121 | 88
  Aspartate aminotransferase increased (grade 3-4) | 3 | 2
  Bilirubin increased (all grades): number analyzed (Participants) | 122 | 88
  Bilirubin increased (all grades) | 13 | 5
  Bilirubin increased (grade 3-4): number analyzed (Participants) | 122 | 89
  Bilirubin increased (grade 3-4) | 1 | 0
  Calcium decreased (all grades): number analyzed (Participants) | 122 | 88
  Calcium decreased (all grades) | 15 | 7
  Calcium decreased (grade 3-4) | 0 | 0
  Calcium increased (all grades): number analyzed (Participants) | 122 | 88
  Calcium increased (all grades) | 1 | 7
  Calcium increased (grade 3-4): number analyzed (Participants) | 125 | 88
  Calcium increased (grade 3-4) | 0 | 3
  Creatinine increased (all grades): number analyzed (Participants) | 122 | 88
  Creatinine increased (all grades) | 73 | 46
  Creatinine increased (grade 3-4): number analyzed (Participants) | 122 | 88
  Creatinine increased (grade 3-4) | 2 | 3
  Glucose decreased (all grades): number analyzed (Participants) | 122 | 88
  Glucose decreased (all grades) | 32 | 26
  Glucose decreased (grade 3-4) | 0 | 0
  Glucose increased (all grades) | NA — Fasting glucose is required for CTCAE grading of hyperglycemia grade 1-2, not grade 3-4. Since fasting glucose was not required for this study, grade 1-2 (glucose-high) could not be determined. Only grade 3-4 was determined. | NA — Fasting glucose is required for CTCAE grading of hyperglycemia grade 1-2, not grade 3-4. Since fasting glucose was not required for this study, grade 1-2 (glucose-high) could not be determined. Only grade 3-4 was determined.
  Glucose increased (grade 3-4): number analyzed (Participants) | 122 | 88
  Glucose increased (grade 3-4) | 10 | 11
  Phosphate decreased (all grades): number analyzed (Participants) | 122 | 88
  Phosphate decreased (all grades) | 42 | 22
  Phosphate decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Phosphate decreased (grade 3-4) | 12 | 6
  Potassium decreased (all grades): number analyzed (Participants) | 122 | 88
  Potassium decreased (all grades) | 25 | 11
  Potassium decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Potassium decreased (grade 3-4) | 2 | 1
  Potassium increased (all grades): number analyzed (Participants) | 122 | 88
  Potassium increased (all grades) | 13 | 17
  Potassium increased (grade 3-4): number analyzed (Participants) | 125 | 88
  Potassium increased (grade 3-4) | 0 | 5
  Sodium decreased (all grades): number analyzed (Participants) | 122 | 88
  Sodium decreased (all grades) | 54 | 28
  Sodium decreased (grade 3-4): number analyzed (Participants) | 122 | 88
  Sodium decreased (grade 3-4) | 10 | 6
  Sodium increased (all grades): number analyzed (Participants) | 122 | 88
  Sodium increased (all grades) | 2 | 1
  Sodium increased (grade 3-4) | 0 | 0
  Urate increased (all grades): number analyzed (Participants) | 122 | 88
  Urate increased (all grades) | 32 | 38
  Urate increased (grade 3-4): number analyzed (Participants) | 122 | 88
  Urate increased (grade 3-4) | 8 | 8
  Amylase increased (all grades): number analyzed (Participants) | 122 | 88
  Amylase increased (all grades) | 20 | 18
  Amylase increased (grade 3-4): number analyzed (Participants) | 122 | 88
  Amylase increased (grade 3-4) | 1 | 3
  Lipase increased (all grades): number analyzed (Participants) | 122 | 88
  Lipase increased (all grades) | 37 | 32
  Lipase increased (grade 3-4): number analyzed (Participants) | 122 | 88
  Lipase increased (grade 3-4) | 12 | 10

9. Secondary Outcome: Incidence of Antitherapeutic Antibody (ATA)
Description: Participants who were tested positive for ATA at any time post-baseline were considered to be transiently positive or persistently positive if >=2 consecutive samples were confirmed as positive.
Time Frame: as for outcome 8
Population: Safety Analysis Set: Participants who received at least one dose of enfortumab vedotin. Here, 'Overall Number of Participants Analyzed' signifies ATA subset (participants with a baseline and at least one post-baseline sample). Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 114 | 81
Participants
  Baseline Negative: number analyzed (Participants) | 112 | 80
  Baseline Negative: Negative post-baseline | 109 | 76
  Baseline Negative: Transiently positive post-baseline | 2 | 3
  Baseline Negative: Persistently positive post-baseline | 1 | 1
  Baseline Positive: number analyzed (Participants) | 2 | 1
  Baseline Positive: Negative post-baseline | 1 | 1
  Baseline Positive: Transiently positive post-baseline | 1 | 0
  Baseline Positive: Persistently positive post-baseline | 0 | 0

10. Secondary Outcome: Disease Control Rate at 16 Weeks (DCR16) Per BICR
Description: Percentage of participants with CR, PR, or stable disease (SD) at Week 16 visit. CR is defined as disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to Week 16
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Percentage of Participants | 50 [41.3 to 59.5] | 58.4 [47.5 to 68.8]

11. Secondary Outcome: DCR16 Per Investigator Assessment
Description: Percentage of participants with CR, PR, or stable disease (SD) at Week 16 visit. CR is defined as disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. The appearance of one or more new lesions is also considered progression. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to Week 16
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Percentage of Participants | 55 [46.0 to 64.1] | 64.0 [53.2 to 73.9]

12. Secondary Outcome: Overall Survival (OS): Primary Analysis
Description: OS is defined as the time from first dose of enfortumab vedotin to death from any cause.
Time Frame: Cohort 1 median follow-up time: 28.4 months [range 0.49, 32.62]; Cohort 2 median follow up time: 13.4 months [range 0.33 to 29.27]
Population: Full analysis set: included all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Months | 12.4 [9.46 to 15.57] | 14.7 [10.51 to 18.20]

13. Secondary Outcome: Number of Participants With Adverse Events (AEs): Primary Analysis
Description: AE=untoward medical occurrence associated with use of study intervention, whether or not considered related. Treatment emergent adverse event (TEAE)=newly occurring/worsening AE after first dose of study treatment, within 30 days after last dose. According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03: Grade(G)3=severe AE, G4=life-threatening, urgent intervention indicated, G5=death related to AE. Participants who discontinued treatment due to treatment related TEAEs captured under TEAEs leading to treatment discontinuation. SAE=event at any dose led to death;life-threatening;required inpatient hospitalization/prolongation of existing hospitalization; persistent/significant disability/incapacity; congenital anomaly/birth defect/ important medical event. Treatment related AEs, SAEs, deaths also included. Treatment relatedness was judged by investigator.
Time Frame: as for outcome 7
Population: Safety Analysis Set: includes all participants who received at least one dose of enfortumab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Participants
  Any treatment-emergent AEs (TEAEs) | 125 | 89
  Treatment-related TEAEs | 117 | 86
  Any grade 3-5 TEAEs | 93 | 62
  Treatment-related grade 3-5 TEAEs | 70 | 49
  Any serious TEAEs | 59 | 35
  Treatment-related serious TEAEs | 24 | 15
  Any TEAEs leading to treatment discontinuation | 21 | 18
  Treatment-related TEAEs leading to treatment discontinuation | 15 | 14
  Any TEAEs leading to death | 7 | 8
  Treatment-related TEAEs leading to death | 0 | 3

14. Secondary Outcome: Pharmacokinetics (PK) Parameter for Enfortumab Vedotin: Maximum Concentration (Cmax) (Serum)
Description: Cmax was derived from the PK blood samples collected. Day 1 data informed by samples collected on Day 1, Day 3, and Day 8. Day 15 data informed by samples collected on Day 15, Day 17, and Day 22.
Time Frame: Collected during cycle 1 and 2 of treatment (each cycle=28 days) at Day 1 pre-dose and end of infusion, Day 3, Day 8 pre-dose and end of infusion, Day 15 pre-dose and end of infusion, Day 17, and Day 22
Population: PK analysis set: all participants who received enfortumab vedotin and from whom at least one blood sample was collected and assayed for enfortumab vedotin, monomethyl auristatin E (MMAE) or total antibody (Tab) concentration. Corresponding records of the time of dosing and sample collection must also be available for all enfortumab vedotin. Here, 'Number Analyzed'= participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (µg/mL)
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 120 | 87
Microgram per milliliter (µg/mL)
  Cycle 1, Day 1 | 26.6 (28.5) | 23.9 (24.4)
  Cycle 1, Day 15: number analyzed (Participants) | 93 | 64
  Cycle 1, Day 15 | 26.0 (28.3) | 21.7 (29.7)
  Cycle 2, Day 1: number analyzed (Participants) | 105 | 73
  Cycle 2, Day 1 | 24.5 (31.4) | 22.0 (24.5)
  Cycle 2, Day 15: number analyzed (Participants) | 95 | 62
  Cycle 2, Day 15 | 26.3 (25.2) | 20.7 (27.4)

15. Secondary Outcome: PK Parameter for Enfortumab Vedotin: Time to Maximum Concentration (Tmax) (Serum)
Description: Tmax was derived from the PK blood samples collected. Day 1 data informed by samples collected on Day 1, Day 3, and Day 8. Day 15 data informed by samples collected on Day 15, Day 17, and Day 22.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Days
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 120 | 87
Days
  Cycle 1, Day 1: number analyzed (Participants) | 119 | 87
  Cycle 1, Day 1 | 0.0278 [0.010 to 0.052] | 0.0264 [0.021 to 0.088]
  Cycle 1, Day 15: number analyzed (Participants) | 92 | 63
  Cycle 1, Day 15 | 0.0285 [0.014 to 0.054] | 0.0264 [0.014 to 0.084]
  Cycle 2, Day 1: number analyzed (Participants) | 104 | 73
  Cycle 2, Day 1 | 0.0264 [0.011 to 0.042] | 0.0264 [0.015 to 0.074]
  Cycle 2, Day 15: number analyzed (Participants) | 94 | 62
  Cycle 2, Day 15 | 0.0285 [0.020 to 0.115] | 0.0257 [0.010 to 0.047]

16. Secondary Outcome: PK Parameter for Enfortumab Vedotin: Area Under Concentration-Time Curve (AUC) (Serum)
Description: AUC was derived from the PK blood samples collected.
Time Frame: AUC0-7 was assessed (in cycles 1 and 2) based on concentration data from Day 1 to Day 8 (pre dose) and AUC0-14 was assessed based on data from D15 (pre dose) to D29 (pre-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 120 | 87
Day*microgram per milliliter
  7-day post-infusion AUC (AUC(d0-7)) - Cycle 1, Day 1: number analyzed (Participants) | 115 | 85
  7-day post-infusion AUC (AUC(d0-7)) - Cycle 1, Day 1 | 34.6 (34.0) | 33.5 (41.4)
  AUC(d0-7) - Cycle 1, Day 8: number analyzed (Participants) | 88 | 63
  AUC(d0-7) - Cycle 1, Day 8 | 31.3 (43.8) | 26.3 (46.0)
  AUC(d0-7) - Cycle 2, Day 1: number analyzed (Participants) | 104 | 72
  AUC(d0-7) - Cycle 2, Day 1 | 36.4 (36.7) | 32.0 (30.0)
  AUC(d0-7) - Cycle 2, Day 8: number analyzed (Participants) | 88 | 56
  AUC(d0-7) - Cycle 2, Day 8 | 35.9 (41.2) | 27.8 (35.8)
  14-day post-infusion AUC (AUC(d0-14)) - Cycle 1, Day 8: number analyzed (Participants) | 85 | 59
  14-day post-infusion AUC (AUC(d0-14)) - Cycle 1, Day 8 | 34.7 (44.7) | 30.9 (47.5)
  AUC(d0-14) - Cycle 2, Day 15: number analyzed (Participants) | 82 | 60
  AUC(d0-14) - Cycle 2, Day 15 | 41.2 (40.4) | 33.1 (36.6)

17. Secondary Outcome: PK Parameter for Free Monomethyl Auristatin E (MMAE): Cmax (Plasma)
Description: as for outcome 14
Time Frame: as for outcome 14
Population: PK analysis set: all participants who received enfortumab vedotin and from whom at least one blood sample was collected and assayed for enfortumab vedotin, MMAE or Tab concentration. Corresponding records of the time of dosing and sample collection must also be available for all enfortumab vedotin. Here, 'Overall Number of Participants Analyzed'=number of participants evaluable for this outcome measure. Here, 'Number Analyzed'= participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 117 | 84
Nanogram per milliliter
  Cycle 1, Day 1 | 3.1 (67.0) | 2.6 (57.8)
  Cycle 1, Day 15: number analyzed (Participants) | 93 | 64
  Cycle 1, Day 15 | 3.9 (64.8) | 3.5 (51.8)
  Cycle 2, Day 1: number analyzed (Participants) | 106 | 72
  Cycle 2, Day 1 | 2.4 (57.4) | 2.2 (60.8)
  Cycle 2, Day 15: number analyzed (Participants) | 90 | 62
  Cycle 2, Day 15 | 3.0 (64.8) | 2.9 (59.9)

18. Secondary Outcome: PK Parameter for Free MMAE: Tmax (Plasma)
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 17
Measure: Median (Full Range); unit: Days
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 117 | 84
Days
  Cycle 1, Day 1 | 1.9 [1 to 5] | 1.9 [1 to 4]
  Cycle 1, Day 15: number analyzed (Participants) | 93 | 64
  Cycle 1, Day 15 | 2.0 [1 to 11] | 1.9 [1 to 9]
  Cycle 2, Day 1: number analyzed (Participants) | 106 | 72
  Cycle 2, Day 1 | 2.0 [1 to 5] | 1.8 [1 to 5]
  Cycle 2, Day 15: number analyzed (Participants) | 90 | 62
  Cycle 2, Day 15 | 1.9 [1 to 9] | 1.9 [1 to 10]

19. Secondary Outcome: PK Parameter for Free MMAE: AUC (Plasma)
Description: AUC was derived from the PK blood samples collected.
Time Frame: as for outcome 16
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*nanogram per milliliter
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 117 | 84
Day*nanogram per milliliter
  7-day post-infusion AUC (AUC(d0-7)) - Cycle 1, Day 1: number analyzed (Participants) | 115 | 84
  7-day post-infusion AUC (AUC(d0-7)) - Cycle 1, Day 1 | 14.1 (81.7) | 13.0 (64.1)
  AUC(d0-7) - Cycle 1, Day 8: number analyzed (Participants) | 88 | 66
  AUC(d0-7) - Cycle 1, Day 8 | 19.1 (79.1) | 18.1 (65.0)
  AUC(d0-7) - Cycle 2, Day 1: number analyzed (Participants) | 104 | 72
  AUC(d0-7) - Cycle 2, Day 1 | 11.3 (58.0) | 10.6 (65.0)
  AUC(d0-7) - Cycle 2, Day 8: number analyzed (Participants) | 88 | 57
  AUC(d0-7) - Cycle 2, Day 8 | 14.9 (64.7) | 15.3 (60.2)
  14-day post-infusion AUC (AUC(d0-14)) - Cycle 1, Day 15: number analyzed (Participants) | 91 | 62
  14-day post-infusion AUC (AUC(d0-14)) - Cycle 1, Day 15 | 25.9 (74.7) | 22.6 (76.4)
  AUC(d0-14) - Cycle 2, Day 15: number analyzed (Participants) | 84 | 63
  AUC(d0-14) - Cycle 2, Day 15 | 19.1 (61.2) | 21.3 (65.0)

20. Secondary Outcome: PK Parameter for Total Antibody (TAb): Cmax (Serum)
Description: as for outcome 14
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 120 | 87
Microgram per milliliter
  Cycle 1, Day 1 | 26.6 (30.4) | 26.4 (23.4)
  Cycle 1, Day 15: number analyzed (Participants) | 93 | 64
  Cycle 1, Day 15 | 30.9 (22.9) | 27.3 (25.7)
  Cycle 2, Day 1: number analyzed (Participants) | 105 | 74
  Cycle 2, Day 1 | 26.2 (30.5) | 26.3 (23.8)
  Cycle 2, Day 15: number analyzed (Participants) | 95 | 62
  Cycle 2, Day 15 | 30.2 (22.7) | 27.1 (28.2)

21. Secondary Outcome: PK Parameter for TAb: Tmax (Serum)
Description: Tmax was derived from the PK blood samples collected. Time of maximum concentration corresponds to the end of infusion sample time. Day 1 data informed by samples collected on Day 1, Day 3, and Day 8. Day 15 data informed by samples collected on Day 15, Day 17, and Day 22.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Days
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 120 | 87
Days
  Cycle 1, Day 1: number analyzed (Participants) | 119 | 87
  Cycle 1, Day 1 | 0.0278 [0.010 to 0.052] | 0.0264 [0.021 to 0.088]
  Cycle 1, Day 15: number analyzed (Participants) | 92 | 63
  Cycle 1, Day 15 | 0.0285 [0.014 to 0.054] | 0.0264 [0.014 to 0.084]
  Cycle 2, Day 1: number analyzed (Participants) | 104 | 74
  Cycle 2, Day 1 | 0.0264 [0.011 to 0.042] | 0.0264 [0.015 to 0.074]
  Cycle 2, Day 15: number analyzed (Participants) | 94 | 62
  Cycle 2, Day 15 | 0.0285 [0.020 to 0.115] | 0.0257 [0.010 to 0.047]

22. Secondary Outcome: PK Parameter for TAb: AUC (Serum)
Description: AUC was derived from the PK blood samples collected.
Time Frame: as for outcome 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 120 | 87
Day*microgram per milliliter
  7-day post-infusion AUC (AUC(d0-7)) - Cycle 1, Day 1: number analyzed (Participants) | 115 | 85
  7-day post-infusion AUC (AUC(d0-7)) - Cycle 1, Day 1 | 63.4 (33.6) | 66.8 (34.3)
  AUC(d0-7) - Cycle 1, Day 8: number analyzed (Participants) | 88 | 63
  AUC(d0-7) - Cycle 1, Day 8 | 77.6 (35.2) | 72.3 (37.9)
  AUC(d0-7) - Cycle 2, Day 1: number analyzed (Participants) | 104 | 72
  AUC(d0-7) - Cycle 2, Day 1 | 73.2 (33.5) | 72.9 (26.4)
  AUC(d0-7) - Cycle 2, Day 8: number analyzed (Participants) | 88 | 56
  AUC(d0-7) - Cycle 2, Day 8 | 87.9 (30.6) | 81.0 (30.9)
  14-day post-infusion AUC (AUC(d0-14)) - Cycle 1, Day 15: number analyzed (Participants) | 93 | 62
  14-day post-infusion AUC (AUC(d0-14)) - Cycle 1, Day 15 | 98.1 (38.8) | 91.1 (40.3)
  AUC(d0-14) - Cycle 2, Day 15: number analyzed (Participants) | 84 | 62
  AUC(d0-14) - Cycle 2, Day 15 | 113.0 (33.8) | 109.7 (41.5)

23. Secondary Outcome: Number of Participants With Adverse Events (AEs): Final Analysis
Description: as for outcome 13
Time Frame: Cohort 1: median treatment duration time: 4.60 months (range 0.5, 43.0); Cohort 2: median treatment duration time: 5.98 months (range 0.3 to 25.8)
Population: Safety Analysis Set: includes all participants who received at least one dose of enfortumab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Participants
  Any treatment-emergent AEs (TEAEs) | 125 | 89
  Treatment-related TEAEs | 117 | 86
  Any grade 3-5 TEAEs | 93 | 62
  Treatment-related grade 3-5 TEAEs | 70 | 49
  Any serious TEAEs | 59 | 35
  Treatment-related serious TEAEs | 24 | 15
  Any TEAEs leading to treatment discontinuation | 22 | 21
  Treatment-related TEAEs leading to treatment discontinuation | 16 | 17
  Any TEAEs leading to death | 7 | 8
  Treatment-related TEAEs leading to death | 0 | 3

24. Secondary Outcome: Overall Survival (OS): Final Analysis
Description: OS is defined as the time from first dose of enfortumab vedotin to death from any cause.
Time Frame: Cohort 1: median follow-up: 61.0 months (range 59.63, 62.36); Cohort 2: median follow-up time: 45.8 months (range 44.91 to 48.95)
Population: Full analysis set: includes all enrolled participants who received at least one dose of enfortumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
Number analyzed (Participants) | 125 | 89
Months | 12.4 [9.46 to 15.57] | 15.6 [11.24 to 20.37]

ADVERSE EVENTS:
Time Frame: Cohort 1: maximum up to 62.36 months of follow-up; Cohort 2: maximum up to 48.95 months of follow-up
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set was evaluated.
Arm/Group | Enfortumab Vedotin - Cohort 1 | Enfortumab Vedotin - Cohort 2
All-Cause Mortality (participants affected / at risk) | 104/125 | 72/89
Serious Adverse Events (participants affected / at risk) | 59/125 | 35/89
Other Adverse Events (participants affected / at risk) | 123/125 | 88/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin - Cohort 1 (N=125) | Enfortumab Vedotin - Cohort 2 (N=89)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 6 (6) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (4)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 9 (10)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (3)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin - Cohort 1 (N=125) | Enfortumab Vedotin - Cohort 2 (N=89)
Neutropenia (Blood and lymphatic system disorders) | 13 (22) | 10 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (11) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 44 (62) | 34 (42)
Palpitations (Cardiac disorders) | 1 (1) | 5 (7)
Tachycardia (Cardiac disorders) | 9 (10) | 1 (1)
Blepharitis (Eye disorders) | 8 (9) | 3 (3)
Dry eye (Eye disorders) | 30 (32) | 17 (19)
Lacrimation increased (Eye disorders) | 21 (25) | 12 (14)
Punctate keratitis (Eye disorders) | 9 (9) | 3 (3)
Vision blurred (Eye disorders) | 20 (25) | 9 (10)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 23 (26) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 5 (7)
Constipation (Gastrointestinal disorders) | 35 (41) | 19 (26)
Diarrhoea (Gastrointestinal disorders) | 52 (73) | 30 (52)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 8 (10)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (9) | 5 (5)
Nausea (Gastrointestinal disorders) | 56 (68) | 26 (35)
Stomatitis (Gastrointestinal disorders) | 10 (11) | 6 (7)
Vomiting (Gastrointestinal disorders) | 24 (36) | 11 (13)
Asthenia (General disorders) | 7 (7) | 7 (15)
Chills (General disorders) | 5 (9) | 7 (8)
Fatigue (General disorders) | 66 (71) | 40 (41)
Gait disturbance (General disorders) | 7 (7) | 9 (9)
Malaise (General disorders) | 10 (10) | 2 (3)
Oedema peripheral (General disorders) | 31 (45) | 20 (22)
Pyrexia (General disorders) | 15 (17) | 14 (16)
Oral candidiasis (Infections and infestations) | 7 (7) | 5 (5)
Urinary tract infection (Infections and infestations) | 18 (23) | 13 (17)
Fall (Injury, poisoning and procedural complications) | 14 (18) | 9 (12)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (5) | 5 (6)
Alanine aminotransferase increased (Investigations) | 15 (16) | 9 (11)
Amylase increased (Investigations) | 13 (17) | 15 (19)
Aspartate aminotransferase increased (Investigations) | 19 (27) | 11 (15)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 1 (1)
Blood creatinine increased (Investigations) | 11 (17) | 5 (10)
Lipase increased (Investigations) | 16 (27) | 9 (15)
Lymphocyte count decreased (Investigations) | 9 (9) | 2 (5)
Weight decreased (Investigations) | 40 (41) | 31 (33)
Decreased appetite (Metabolism and nutrition disorders) | 64 (81) | 35 (43)
Dehydration (Metabolism and nutrition disorders) | 12 (14) | 10 (11)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (20) | 12 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 8 (14) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (20) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (17) | 9 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (12) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (16) | 10 (10)
Dizziness (Nervous system disorders) | 20 (23) | 10 (12)
Dysgeusia (Nervous system disorders) | 49 (53) | 27 (28)
Headache (Nervous system disorders) | 6 (6) | 5 (6)
Paraesthesia (Nervous system disorders) | 4 (4) | 6 (7)
Peripheral motor neuropathy (Nervous system disorders) | 14 (16) | 9 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 54 (59) | 47 (53)
Anxiety (Psychiatric disorders) | 4 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 18 (18) | 13 (13)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 6 (6)
Dysuria (Renal and urinary disorders) | 6 (6) | 5 (6)
Haematuria (Renal and urinary disorders) | 10 (13) | 10 (11)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 12 (15)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 14 (16)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 64 (67) | 48 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 35 (38) | 18 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (41) | 31 (37)
Rash erythematous (Skin and subcutaneous tissue disorders) | 15 (16) | 6 (10)
Rash macular (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 (45) | 28 (40)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7 (10) | 3 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 13 (14) | 4 (4)
Hypertension (Vascular disorders) | 7 (12) | 4 (5)
Hypotension (Vascular disorders) | 9 (10) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT03219333/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT03219333/SAP_001.pdf